CLINICAL TRIAL: NCT02117609
Title: Effet d'Une supplémentation Avec Une Nouvelle préparation hyperprotéinée et Hypercalorique Sur l'évolution Des paramètres Fonctionnels, Nutritionnels et Cognitifs Chez la Personne âgée en Institution
Brief Title: Effect of a New High-protein Oral Supplement on Functional Parameters in Patients in Nursing Homes
Acronym: PRESAGE-T2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lactalis (Industry)
Collaborators: University Hospital, Toulouse (Other); University of Lille Nord de France (Other); National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LRD-2011-PRESAGE; ANR ALIA2010-01306 Presage (Other Grant/Funding Number: National Research Organization, France)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Malnutrition
Keywords: Elderly; Nursing home; Functional impairment; High-protein oral supplement
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- New DELICAL formula (Experimental): New high-protein oral nutrient supplement
  Interventions: Dietary Supplement: New DELICAL formula
- Standard DELICAL formula (Active Comparator): Standard isoenergetic isoprotein formula
  Interventions: Dietary Supplement: Standard DELICAL formula

INTERVENTIONS:
Dietary Supplement: New DELICAL formula — 3 months with the option of continuing until 6 months.
  Arms: New DELICAL formula
Dietary Supplement: Standard DELICAL formula — 3 months with the option of continuing until 6 months.
  Arms: Standard DELICAL formula

SUMMARY:
The objective of this study is to determine whether a supplementation with a new high-protein oral supplement can improve the evolution of functional parameters in elderly patients in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged more than 60 years old
* Living in a nursing home for at least 2 months
* Malnourished or at risk of malnutrition (MNA<23.5 or BMI<24 or albumin<35 g/l or weight loss of more than 5 kg in the last 6 months)
* Without dementia or with moderate dementia (MMSE > or =10/30)
* Able to walk without human assistance (technical assistance allowed)
* No vitamin D supplementation
* Able to follow the study procedures and agreed to consume oral supplement

Exclusion Criteria:

* Severe dementia (MMSE < 10/30)
* Enteral nutrition
* Severe renal or hepatic impairment
* Cancer with chemotherapy
* Uncontrolled diabetes
* Lactose intolerance
* Cow's milk protein allergy

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 4-meter walking speed | After 3 months and 6 months

SECONDARY OUTCOMES:
Change from baseline in grip strength | After 3 months and 6 months
Change from baseline in ADL (Activities Daily Living) score | After 3 months and 6 months
Change from baseline in Geriatric Depression Scale | After 3 months and 6 months
Change from baseline in quality of life (QOL-AD) | After 3 months and 6 months
Frequency of pathologic adverse events (disease, acute infection, falls, hospitalization) | During the 3 months and/or 6 months of consumption
Change from baseline in body composition measured by bioelectrical impedence analysis (BIA) | After 3 months and 6 months
Change from baseline in nutritional status (Mini Nutritional Assessment) | After 3 months and 6 months
Changes from baseline in blood parameters | After 3 months and 6 months
  Inflammation markers (TNFalpha, TNF-R1, TNF-R2, IL 15), Fatty acid composition of red blood cell membranes, Fibrinogen, CRP, albumin, prealbumin, orosomucoid, IGF-1, cystein, glutathione peroxidase, oxidized and reduced glutathione

CONTACTS AND LOCATIONS:
Overall Officials: Yves Rolland, Pr, Principal Investigator — University Hospital, Toulouse; Cécile Bonhomme, PhD, Study Director — Lactalis Nutrition Santé; David Seguy, Dr, Study Chair — U995, Université Lille Nord France; Charlotte Baudry, PhD, Study Chair — Lactalis Recherche et Développement
Locations (1):
- Nursing homes - Région Midi-Pyrénées, Toulouse, France